CLINICAL TRIAL: NCT02565056
Title: Acceptance and Commitment Therapy Self-help Intervention for Depression in Haemodialysis Patients: A Feasibility Randomised Controlled Trial
Brief Title: Feasibility RCT of ACT Self-help for Depression in Haemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lincoln (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, William Vogt, Trainee Clinical Psychologist, University of Lincoln
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 156756
Record Dates: First submitted 2015-09-23; First posted 2015-10-01 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: End-stage Renal Disease; Depression
Keywords: Acceptance and Commitment Therapy
MeSH Terms: conditions — Kidney Failure, Chronic; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-help (Active Comparator): Self-help book completed over 6 weeks with up to 30 minutes of telephone support per week.
  Interventions: Other: Self help book + telephone support
- Treatment as usual (No Intervention): Treatment as usual.

INTERVENTIONS:
Other: Self help book + telephone support — Self-help book based upon principles of Acceptance and Commitment Therapy
  Arms: Self-help

SUMMARY:
The purpose of this study is to assess the feasibility of conducting a trial to evaluate a self-help treatment for depression in people with end-stage renal disease.

DETAILED DESCRIPTION:
Chronic Kidney Disease (CKD) is a long-term condition in which the function of the kidneys - to filter out waste products from the blood - slowly declines. When renal function becomes sufficiently low it is described as End Stage Renal Disease (ESRD) and renal replacement therapy (RRT) is likely to be needed to prolong life. The most common type of RRT is haemodialysis, in which the patient's blood is filtered through a machine.

It is estimated that depression is experienced by 20-40% of people with ESRD. Depression not only affects the quality of life of individuals with ESRD but is also associated with higher rates of hospitalisation and poorer physical health outcomes.

Acceptance and Commitment Therapy (ACT) has been found to be an effective treatment for depression and has been used successfully as a self-help treatment. However, no study has examined the effectiveness of an ACT self-help treatment for depression in ESRD. This study aims to assess the feasibility of conducting such a study and will look at suitability of recruitment, assessment methods and the acceptability of the self-help treatment, as well as helping to calculate the number of people needed for a definitive study.

Haemodialysis patients receiving dialysis through an NHS renal service will be invited to participate. To participate they will be consenting, over 18 years of age and experiencing depressive symptoms at a clinical level. Those eligible will be randomly assigned into one of two conditions; a control condition receiving treatment as usual (TAU), and an intervention condition receiving TAU alongside an ACT self-help manual with weekly telephone support. The manual will be completed over six weeks. Both groups will be asked to complete questionnaires prior to intervention and 2 and 4 months post-intervention. Participants from each condition will be asked to participate in interviews to explore their experiences of taking part.

ELIGIBILITY:
Inclusion Criteria:

* undergoing haemodialysis treatment at one of three identified units
* receiving haemodialysis treatment for more than 6 months
* moderate depression (as indicated by the PHQ-9)

Exclusion Criteria:

* receiving concurrent psychological treatment
* lacking mental capacity to consent due to cognitive impairment
* inadequate reading ability (indicated by inability to complete PHQ-9 screening measure)
* visual or hearing impairment that would prevent completion of the self-help book or engagement in telephone calls

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire (PHQ-9) at 2 and 4 months | Baseline; 2 months; 4 months
  Validated self-report questionnaire assessing symptoms of depression

SECONDARY OUTCOMES:
Change in EQ-5D-5L at 2 and 4 months | Baseline; 2 months; 4 months
  Validated self-report questionnaire assessing health-related quality of life
Change in Acceptance and Action Questionnaire - 2 (AAQ-2) at 2 and 4 months | Baseline; 2 months; 4 months
  Validated self-report questionnaire assessing psychological flexibility
Change in Valued Living Questionnaire (VLQ) at 2 and 4 months | Baseline; 2 months; 4 months
  Validated self-report questionnaire assessing the extent to which individuals live consistently with their identified values

CONTACTS AND LOCATIONS:
Overall Officials: William Vogt, MSc, BSc, Principal Investigator — University of Lincoln
Locations (3):
- United Kingdom (3):
  - Shipley Dialysis Unit, Ilkeston Community Hospital, Ilkeston, Derbyshire
  - Mike Cassidy Dialysis Unit, Kings Mill Hospital, Mansfield, Nottinghamshire
  - Main Dialysis Unit & Centenary Dialysis Unit (same site), City Hospital, Nottingham, Nottinghamshire